CLINICAL TRIAL: NCT01793207
Title: Peripheral Blood DNA Methylation Markers for the Early Detection of Colorectal Carcinoma in the Egyptian Population
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); science and technology development fund, Egypt (Unknown)
Responsible Party: Principal Investigator, Hany Shehab, Dr., Cairo University
Other Study IDs: CRCS001; 3023 (Other: Egyptian Science and Technological Development Fund)
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Colorectal Neoplasms; Adenoma; Colorectal Tumors
MeSH Terms: conditions — Colorectal Neoplasms; Adenoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 10cc blood sample and tissue biopsies from colorectal lesions when present.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Normal: Subjects who had a normal colonoscopic examination (No polyps, masses or any evidence of colorectal neoplasia)
- colorectal cancer: Patients with endoscopic and histopathological evidence of colorectal cancer
- Adenoma: Patients with colorectal adenomas only detected on colonoscopy
- Hyperplastic polyps: Patients with hyperplastic polyps detected on colonoscopy.

SUMMARY:
The incidence of colorectal cancer (CRC) is on the rise on a global scale. The number of cancer-related deaths related to CRC is also rising to an alarming level. This picture is similarly seen in Egypt where the incidence of colorectal carcinoma is increasing annually, moreover, CRC in Egypt exhibits an alarming characteristic which is the affection of much younger patients than their counterparts worldwide. Fortunately, the early detection of CRC and its precursor (adenoma) has been shown to markedly decrease morbidity and mortality related to this tumor, this has prompted the development of robust screening programs for CRC in several western countries. The implementation of a CRC screening program in Egypt has been hampered by the low compliance of the patients and the relatively high cost of colonoscopy. There is a need for an affordable, non-invasive, simple, accurate and socially accepted screening test to allow such a program to succeed in Egypt. Recent studies have shown that DNA is the future target of screening tests for several malignancies. Particularly for CRC a few preliminary studies have shown encouraging results with separate DNA methylation markers both in blood and stool. In our efforts to develop a screening test with the criteria stated above, the investigators have decided to join the forces of 2 of the largest medical centers in Egypt and the middle-east: Kasr-Alaini hospital and the National cancer institute (NCI). The investigators plan to test a panel of 7 DNA methylation markers in peripheral blood for their performance as an early marker for CRC and colorectal adenomas. Data from this study will pave the way for the development of a screening test for CRC "tailored" to the Egyptian population, moreover, it will supply essential data about the genetic alterations occurring in CRC in Egyptian patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing colonoscopy as part of their clinical care or part of screening program.
* Complete endoscopic examination (up to the caecum)
* Adequate colonic preparation

Exclusion Criteria:

* - Incomplete colonoscopic examination due to technical causes e.g. difficult colonoscopy, patient intolerance (N.B. a neoplastic mass causing lumen stenosis will not be excluded.)
* Poor colonic preparation obscuring adequate mucosal examination.
* Patients who have received any treatment for CRC and/or adenomas.
* Patients with known malignancy elsewhere (i.e. non-colorectal malignancy)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients refered to Kasr-Alaini endoscopy unit and National cancer institute endoscopy department for colonoscopy.
Sampling Method: Probability Sample
Enrollment: 316 (Actual)
Dates: Start 2012-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Methylation markers present in peripheral blood of patients with colorectal cancer(Sept 9, CDKN2B-p15, CDH4, SFRP2, ALX4, Neurog1 and CDH13)in comparison to their presence in other subjects | 16 months

SECONDARY OUTCOMES:
Methylation markers present in peripheral blood of patients with colorectal adenomas (Sept 9, CDKN2B-p15, CDH4, SFRP2, ALX4, Neurog1 and CDH13)in comparison to their presence in other subjects | 16 months
Methylation markers present in peripheral blood of patients with hyperplastic polyps(Sept 9, CDKN2B-p15, CDH4, SFRP2, ALX4, Neurog1 and CDH13)in comparison to their presence in other subjects | 16 months

CONTACTS AND LOCATIONS:
Overall Officials: Hany M Shehab, MD, MRCP, Principal Investigator — Cairo University
Locations (2):
- Egypt (2):
  - Kar-Alaini hospital (Cairo Univeristy hospital), Cairo
  - National cancer institute, Cairo